CLINICAL TRIAL: NCT00807274
Title: Prospective Evaluation of Renal Function in Adults With Congenital Heart Disease.
Brief Title: Renal Function in Adults With Congenital Heart Disease.
Status: Withdrawn | Type: Observational
Why Stopped: Alternative trial planned
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Dr Lorna Swan, Royal Brompton Hospital
Other Study IDs: 06/Q0404/75
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Last update posted 2009-09-25 (Estimated); Status verified 2009-09

CONDITIONS: Cardiovascular Abnormalities; Kidney Failure
Keywords: Adult congenital heart disease; Heart failure; Renal failure; Proteinuria
MeSH Terms: conditions — Cardiovascular Abnormalities; Renal Insufficiency; Heart Defects, Congenital; Heart Failure; Proteinuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, serum and urine samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Impaired kidney function is associated with a poor outcome in patients with heart failure but it is not known of this is the case for patients who have been born with their heart condition (congenital heart disease). This study aims to investigate how frequently patients with congenital heart disease have kidney disease and whither this does have an impact on their outcome. The hypothesis is that kidney dysfunction will be common in these patients and may have an impact on long-term health and life-expectancy.

DETAILED DESCRIPTION:
Renal dysfunction is a recognised independent prognosticator in patients with chronic heart failure. Indeed it has been suggested that the clinical impact of renal dysfunction may be greater than that of left ventricular ejection fraction per se.

The role of renal function has also been investigated in small sub-groups of patients with adult congenital heart disease (ACHD) for example peri-operatively. It is not however known if renal dysfunction has the same prevalence and significance as when present to patient with acquired heart failure. The hypothesis of the study is that renal dysfunction, both overt and sub-clinical, will be commonly detected in patients with congenital heart disease. The study proposes that renal dysfunction will be associated with hospitalisation for heart failure and fluid overload and will also identify patients at an increased risk of worsening clinical status.

Comparisons: Baseline renal function (creatinine, glomerular filtration rate by equation and clearance testing), quantification of urinalysis, baseline neurohormones. Follow-up data regarding clinical endpoints including new arrhythmia, functional deterioration, and hospitalisation.

ELIGIBILITY:
Inclusion Criteria:

* The ability to give informed consent
* Age >18 years
* Congenital heart disease being treated as an outpatient

Exclusion criteria:

* Pregnancy
* Renal failure requiring renal-replacement therapy
* Known diabetes
* Shellfish, iodine, or significant drug allergy (sub-study only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stable adult patients with congenital heart disease
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2008-09; Study Completion 2010-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Lorna Swan, MRCP MD, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Adult Congenital Heart Disease Unit, Royal Brompton Hospital, London, London, United Kingdom